CLINICAL TRIAL: NCT02939092
Title: The Effect of Mouthwash Containing Pomegranate Peel Extract and Chlorhexidine Mouthwash on Bleeding on Brushing Among a Group of Egyptian Children With Full Permanent Dentition, Randomized Controlled Trial
Brief Title: The Effect of Mouthwash Containing Pomegranate Peel Extract and Chlorhexidine Mouthwash on Bleeding on Brushing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Heba Moahmed Fouad, Principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CairoE
Record Dates: First submitted 2016-10-11; First posted 2016-10-19 (Estimated); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Gingival Bleeding
Keywords: Gingival Bleeding on probing
MeSH Terms: conditions — Gingival Hemorrhage | interventions — Chlorhexidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pomegranate peel extract (Experimental): Pomegranate is antimicrobial, anti inflammatory and antioxidant
  Interventions: Drug: Pomegranates peel extract
- Chlorhexidine (Active Comparator): Chlorhexidine mouthwash is antiplaque treatment and effective against gingivitis
  Interventions: Drug: Chlorhexidine

INTERVENTIONS:
Drug: Pomegranates peel extract — Pomegranate is antimicrobial
  Arms: Pomegranate peel extract
Drug: Chlorhexidine — Chlorhexidine mouthwash is antiplaque agent
  Arms: Chlorhexidine

SUMMARY:
To evaluate the clinical effectiveness of mouthwash containing pomegranate peel extract and chlorhexidine mouthwash on bleeding on brushing and counting of streptococcus mutans among a group of Egyptian children with permanent dentition.

DETAILED DESCRIPTION:
To evaluate the clinical effectiveness of mouthwash containing pomegranate peel extract and chlorhexidine mouthwash on bleeding on brushing and counting of streptococcus mutans among a group of Egyptian children with permanent dentition.

PICO:

Population (P): Children with full permanent dentition. Intervention (I): Pomegranates peel extract. Comparator (C): Chlorhexidine.

Outcome(O):

Primary outcome: Bleeding on brushing, criteria:Asking patient, unit:Binary. Secondary outcome:Counting streptococcus mutans, criteria: Agar plate, unit: CFUs/mL

ELIGIBILITY:
Inclusion Criteria:

* children aged 12-15 years old.
* Cooperative children.
* Both genders.
* Medically free.

Exclusion Criteria:

* Children undergoing orthodontic treatment.
* Children using any other oral hygiene aid other than routine teeth brushing.
* Children with known history of allergy to any mouth rinse or drug.
* Parents unable to give informed consent.

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2018-01 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Bleeding on brushing, Measurement: asking patient , Unit: Binary | 2 weeks

SECONDARY OUTCOMES:
Counting streptococcus mutans, Measurement: Agar plate, Unit: CFUs/mL | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Salah El Behery, Professor, Study Director — Cairo University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Howell AB, D'Souza DH. The pomegranate: effects on bacteria and viruses that influence human health. Evid Based Complement Alternat Med. 2013;2013:606212. doi: 10.1155/2013/606212. Epub 2013 May 20. PMID 23762148
- [Background] Umar D, Dilshad B, Farhan M, Ali A, Baroudi K. The effect of pomegranate mouthrinse on Streptococcus mutans count and salivary pH: An in vivo study. J Adv Pharm Technol Res. 2016 Jan-Mar;7(1):13-6. doi: 10.4103/2231-4040.173266. PMID 26955605
- [Background] Tulsani SG, Chikkanarasaiah N, Siddaiah SB, Krishnamurthy NH. The effect of Propolis and Xylitol chewing gums on salivary Streptococcus mutans count: a clinical trial. Indian J Dent Res. 2014 Nov-Dec;25(6):737-41. doi: 10.4103/0970-9290.152182. PMID 25728105
- [Background] Ajdic D, McShan WM, McLaughlin RE, Savic G, Chang J, Carson MB, Primeaux C, Tian R, Kenton S, Jia H, Lin S, Qian Y, Li S, Zhu H, Najar F, Lai H, White J, Roe BA, Ferretti JJ. Genome sequence of Streptococcus mutans UA159, a cariogenic dental pathogen. Proc Natl Acad Sci U S A. 2002 Oct 29;99(22):14434-9. doi: 10.1073/pnas.172501299. Epub 2002 Oct 23. PMID 12397186
- [Background] Filoche SK, Soma K, Sissons CH. Antimicrobial effects of essential oils in combination with chlorhexidine digluconate. Oral Microbiol Immunol. 2005 Aug;20(4):221-5. doi: 10.1111/j.1399-302X.2005.00216.x. PMID 15943766
- [Background] Zarfeshany A, Asgary S, Javanmard SH. Potent health effects of pomegranate. Adv Biomed Res. 2014 Mar 25;3:100. doi: 10.4103/2277-9175.129371. eCollection 2014. PMID 24800189
- See also: Related Info — http://doi.org/10.4103/2231-4040.173266
- See also: Related Info — http://www.ijdr.in/text.asp?2014/25/6/737/152182
- See also: Related Info — http://doi.org/10.4103/2277-9175.129371